CLINICAL TRIAL: NCT02853188
Title: Does the Measure of the Plasma Tissue Factor Allow to Predict a Venous Thromboembolism Episode for Patients Presenting a Primitive Lung Cancer?
Brief Title: Measure of Plasma Tissue Factor to Predict a Venous Thromboembolism in Primitive Cancer of Lung
Acronym: FT-KBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014/21; 2014-A00881-46 (Other: ANSM)
Record Dates: First submitted 2016-07-27; First posted 2016-08-02 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Cancer of Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cancer of lung (Experimental)
  Interventions: Other: venous thromboembolism

INTERVENTIONS:
Other: venous thromboembolism

SUMMARY:
The aim of the study is to evaluate if the plasma activity of the tissue factor at the time of the diagnosis of a lung cancer, before any treatment, or after the treatment of induction (surgery or two first cures of chemotherapy), can be a predictive factor of venous thromboembolism disease in the year which follows the diagnosis, independently of the other parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients of more than 18 years old
* Patients with cancer of lung diagnosis carried for less than 2 months and which were not handled yet, either by surgery or by chemotherapy, or by radiotherapy
* Patients whose life expectancy is considered 3-month-old a superior
* Patients having given writed consent
* Patients affiliated to a national insurance scheme or benefiting from such a diet
* Patients having received a treatment (processing) anticoagulating in preventive dose if this treatment was stopped at least 3 days before the 1st taking or patients not receiving an anticoagulating treatment (in case of curative treatment, the latter was before arrested at least 3 months

Exclusion Criteria:

* Patients having a hepatic disease with coagulation disorders
* Patients under anticoagulants with dose guardian in 3 months preceding the study or presenting an active infection
* Patients having a history of other cancer considered as cured and diagnosed for less than 5 years (with the exception of the patients operated for an in situ carcinoma of the neck of the womb or the patients having undergone the excision of a squamous-cell carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism occurence | 2 years
Tissue factor | 2 years
  Tissue factor is measured by kinetic-chromogenic assay

CONTACTS AND LOCATIONS:
Overall Officials: Marc VASSE, PhD, Study Director — Hopitak Foch
Locations (5):
- France (5):
  - Centre hospitalier intercommunal de Créteil, Créteil
  - Centre hospitalier de Versailles, Le Chesnay
  - : Institut Mutualiste Montsouris, Paris
  - AP-HP Hôpital Européen Georges Pompidou, Paris
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No